CLINICAL TRIAL: NCT05159102
Title: Fit Families Program: Fundamental Motor Skill Intervention in Children With Autism Spectrum Disorders and Their Parents
Brief Title: Fit Families Program for Families of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1256 New Cohort; A176000 (Other: UW Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW Madison)
Record Dates: First submitted 2021-10-11; First posted 2021-12-15 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Workshop group (Experimental): Participants in the workshop group will be offered four one-day workshops (3-hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) Sports (during intervention)-[Parents and Children-Workshop Group]. These workshops will be offered in person. In addition to the workshops, this group and the home-based group will receive information (activity booklets via the Fit Families App) and physical education (physical activity)-related equipment.
  Interventions: Other: 12-week FMS Intervention; Behavioral: Physical Activities & Activity Booklets (via FitFamilies app)
- Home-based group (Experimental): Participants in the home-based group will not participate in the four half-day workshops (face to face), but they will receive the same information remotely (workshop content) and will have access to the activity booklets (via the App) and physical activity equipment as the workshop group (during intervention)-[Parents and Children-Home Group].
  Interventions: Other: 12-week FMS Intervention; Behavioral: Physical Activities & Activity Booklets (via FitFamilies app)
- wait-listed home-based group (Other): Wait-list home-based group will serve as the control group (during intervention)-[Parents and Children-Control Group]. This group will be instructed to continue their typical routines and activities for the duration of the intervention. They will be asked to attend the pre and posttest, as well as a follow up three weeks after the completion of the 12-week period. Immediately following the follow-up test, participants in the wait-list home-based group will be offered the home-based program (e.g., receiving the same intervention protocol and materials (physical education equipment and lesson plans/workbook) following all procedures as described for that group previously.
  Interventions: Behavioral: Physical Activities & Activity Booklets (via FitFamilies app)

INTERVENTIONS:
Other: 12-week FMS Intervention — 4 sessions, no more than 3 hours per session covering 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) and Sports (during intervention)
  Arms: Home-based group; Workshop group
Behavioral: Physical Activities & Activity Booklets (via FitFamilies app) — expected to engage in physical activity at least 3 hours per week, parent workshops provide them with resources to engage in Physical activity
  Other Names: Parent workshops

SUMMARY:
The purpose of the study is twofold. First, to identify the effect of a 12-week fundamental motor skills (FMS) (e.g., throwing, catching, running) intervention on the active participation in physical recreation activities as well as a variety of other factors (child behaviors, communication, and adaptive skills). Second, to identify patterns, benefits, constraints, and strategies to active participation in physical recreation activities among families of children with autism spectrum disorders (ASD) (pre-post) through in-person or via phone interviews with parents and children with ASD. Participants will be randomly assigned to one of three protocols: 1) Workshop group, 2) Home-based group, and 3) Wait-listed home-based group. Participants in all groups will receive an activity booklet (in the form of an App) and physical education-related activity items (e.g., ball, hoop).

The investigators hypothesize that both the workshop and home-based groups will improve in all measures from pre to post compared to the wait-list control group. The investigators want to determine if the differences in the workshop and home-based groups differ significantly or are equitable in terms of gains in all areas.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three groups (e.g., workshop, home-based, or control group) (pre-intervention)- [Parents and Children]. Group assignment will occur once pre-measurements/interviews data has been collected. Each family will be notified via email or phone which group they have been assigned (e.g., workshop, home-based, or control group) families within one week of the initial visit.

* Note: Depending on the COVID situation and if necessary, some components of the program from in-person may be moved to virtual learning. Thus, instead of having three groups, there will be two groups. One online and a wait-listed control group. Parents will be notified about these changes verbally and/or via email.

Parents and children assigned to the workshop group will be asked to participate in a 12 week FMS intervention (no more than three hours per session) and would be expected to engage in the physical activities provided (at least 3 hours per week). The homegroup would also be expected to engage in the physical activities provided (at least 3 hours per week). Instead of attending the in-person workshop, these participants will be able to attend the workshops remotely on zoom. A zoom link will be provided to the families the day before the workshop so they can join the event. The waitlist control group will continue the normal activities and would not be provided with physical activities or be expected to participate in any physical activities. Prior to the first workshop, parents in the home-based and the workshop group will be provided with the dates they should come to the Medical Science Building or Schools in the Madison School District (depending on availability) to collect the equipment and activity booklets (via the APP). Also, the investigators will indicate to parents in the workshop group that they will receive an email from the study team with additional information about the workshop and how to prepare for it. Parents in the wait-list control group will be notified of the tentative dates for the post and follow-up data collection, and a tentative time they will be able to benefit from the program (most likely fall 2021- spring 2022).

Participants in the workshop group will be offered four one-day workshops (3-hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) Sports (during intervention)-[Parents and Children-Workshop Group]. These workshops will be offered in person. For the homegroup, these workshops will be offered online via Zoom. In addition to the workshops, this group and the home-based group will receive information (activity booklets via the Fit Families App) and physical education (physical activity)-related equipment. These activities are very similar to activities children will do during their physical education classes. Each face-to-face workshop is divided into two sessions. In the first session, parents attend a seminar and learn techniques and routines integrating the workshop topic into PA experiences that they will practice with their children in the second session. During the first session, children participate in physical activities led by trained staff, separate from their parents. After a mid-morning break, the parents and children are reunited and the parents practice the activities they learned with their children, under guided supervision and modeling from staff. This second session with support serves as a means of reinforcing recently presented skills and individualizing the instruction to the needs of each child and family.

Families in this study (both groups) will be part of a private Facebook page in which they can ask questions or share information related to the program. In addition, study staff will be sharing teaching tips and answer questions families may have using the Facebook page. Making Facebook as an alternative and easy option for these families. WebEx or Zoom requires that users download an application into their computers or devices. The online portions of the program will be either pre-recorded or distributed live to each family (depending on conversations with Help Desk). Families will need to have access to internet services either through their phones or personal computers or devices. Note: To study team knowledge, these families have already access to the internet or mobile technology because, in order to participate in the study, they are required to complete an online application. The online session will not include the practice component in which parents practice the skills learned with their children. In turn, the investigators will ask families to share a video on the private Facebook page of them with their children practicing the skills. Parents will be given the option to send these videos privately to the study team or if they prefer, they can share their videos with the participants in the study (similar to what they will be doing in the face-to-face interactions). Each family will receive the equipment related to the workshop 2 days prior to the workshop. The study team will coordinate the pick-up time and location with each family. The duration of the online workshop is equivalent to face-to-face interactions (approximately 2 and a half hours). Breaks will be provided as requested by the participants.

* Note: depending on the COVID pandemic and university regulations in terms of in-person contact, the study team may mail the equipment to the participant utilizing a local company (e.g., UPS, etc).

Participants in the home-based group will not participate in the four half-day workshops (face to face), but they will receive the same information remotely (workshop content) and will have access to the activity booklets (via the App) and physical activity equipment as the workshop group (during intervention)-[Parents and Children-Home Group]. These two groups (workshop group and home-based group) will be part of two separate closed Facebook page in which only participants enrolled in the page will have access to the content. The purpose of this Facebook page is to have a place in which parents can share information or ask questions to other parents about the physical activities and the physical education-related equipment they will receive. The study team will have access to the Facebook page to monitor the page and provide feedback when needed.

Participants in the workshop and home-based group will be contacted by members of the research team on a weekly basis (during the length of the program) by phone or via email (depending on parental preferences) to follow up on the progress of each family and to clarify questions they may have regarding the information provided. In addition, participants in both intervention groups will receive weekly motivational text messages encouraging them to continue practicing the activities.

Note: The study team will be taking photographs and videos of participants (parents and children) during the workshops at the Medical Science Building or Schools in the Madison School District (depending on availability) and/or during data collection. The photos and the videos will be used for educational purposes.

The third group (wait-list home-based group) will serve as the control group (during intervention)-[Parents and Children-Control Group]. This group will be instructed to continue their typical routines and activities for the duration of the intervention. They will be asked to attend the pre and post-test, as well as a follow-up three weeks after the completion of the 12-week period. Immediately following the follow-up test, participants in the wait-list home-based group will be offered the home-based program (e.g., receiving the same intervention protocol and materials (physical education equipment and lesson plans/workbook) following all procedures as described for that group previously.

The initial cohort of this study was registered to NCT04612647.

ELIGIBILITY:
Parents (one per family) and children with ASD ages 4 to 11 will be included (recruited as a dyad).

Inclusion Criteria:

* ASD must be the primary disability of the child
* Children will be considered to have ASD if they score above the clinical cutoff or 15 on both the lifetime and current versions of the SCQ. Diagnostic severity of ASD will not be a factor in recruitment.
* Children must be able to participate in the program activities.
* Children must be ambulatory and able to follow verbal or picture directions with support
* Children with significant communication needs will still be considered for the study
* No age restriction for adults (parents of children with ASD)
* Parents should be ambulatory and not have any restriction to do physical activity

Exclusion Criteria:

* Parents of children with other primary disabilities, or parents who do not have children with ASD will be excluded.
* Participants cannot exhibit aggressive behavior
* Children who are non-ambulatory, or participants (children) with significant behavioral or sensory impairments will also be excluded based on application information, including existing behavior intervention plans and existing school information

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Development as Measured by TGMD-3 | Baseline, 3 week post intervention (15 weeks)
  The Test of Gross Motor Development - second edition (TGMD-3) is a measure of fundamental motor skills. The total possible range of scores is 47-158, where higher scores are indicative of improved gross motor development.
Change in qualitative perceptions of the participants as measured via semi-structured interview. | baseline (approximately 2 weeks prior to intervention), post intervention (12 weeks), follow up (24 weeks)
  Children will participate in one-on-one semi-structured interviews with the research team to explore their perception regarding communication strategies (between parent and child), patterns of physical recreation, perceived benefits, and constraints.
Change in Social Communication Questionnaire (SCQ) | baseline (approximately 2 weeks prior to intervention), post intervention (12 weeks)
  The SCQ is a 40-item survey where each question is a 'yes' or 'no' answer. The total possible range of scores is 0-39 (verbal children) or 0-33 (non-verbal children) with higher scores indicative of greater frequency of symptoms.
Change in Parenting Stress Index (PSI)- Short form | Baseline, 3 week post intervention (15 weeks)
  The Parenting Stress Index (PSI)- short form is used to measure the relative stress in the parent-child relationship. Parents complete the PSI Short Form test sheet including basic demographic information on the top of the questionnaire first. For most items, parents should respond by circling SA (strongly agree), A (agree), NS (not sure), D (disagree), SD (strongly disagree). Higher raw scores indicate higher levels of stress. Percentile scores that fall between 15 and 80 are considered typical.
Change in Sensory Profile (Dunn 1999) | Baseline, 3 weeks post intervention (15 weeks)
  The Sensory Proﬁle (Dunn, 1999) is designed to function as a part of a broader assessment of a child's functioning, which may include other observations, history, and diagnostic tests. The parent/caregiver reports the frequency of the behaviors in question, utilizing a Likert scale of always, frequently, occasionally, sometimes, and never. The Sensory Proﬁle consists of 125 items grouped into three main sections: sensory processing, modulation, and behavioral and emotional responses.
Change in the Behavioral Assessment System for Children (BASC-III) (Reynolds & Kamphaus, 2015) | Baseline, 3 week post intervention (15 weeks)
  To evaluate social behavior, problem behavior, and emotionality of the child. The narrative and scale classifications in this report are based on T scores obtained using norms. Scale scores in the Clinically Significant range suggest a high level of maladjustment. Scores in the At-Risk range may identify a significant problem that may not be severe enough to require formal treatment or may identify the potential of developing a problem that needs careful monitoring.
Change in Adaptive Behavior Assessment System (ABAS-3) | Baseline, 3 week post intervention (15 weeks)
  To evaluate adaptive behavior skills of the child. The ABAS-3 covers three broad adaptive domains: Conceptual, Social, and Practical. Within these domains, it assesses 11 adaptive skill areas (each form assesses 9 or 10 skill areas based on age range). Items focus on practical, everyday activities required to function, meet environmental demands, care for oneself, and interact with others effectively and independently. On a four-point response scale, raters indicate whether the individual can perform each activity, and if so, how frequently they perform it when needed.
Change in Physical Activity Questionnaire | Baseline, weekly throughout the 12 weeks, post intervention (15 weeks)
  Parents will be asked to complete a weekly Qualtrics survey inquiring about the type of activities and time they spend participating in those activities. In this survey, parents will comment on the FMS strategies they used or did not use during the week(s).

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Columna, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Prieto LA, Meera B, Barry A, Swarup G, Asmus J, Ku B, Roth K, Foley JT, Columna L. A randomized parent-mediated physical activity intervention for autistic children. Autism Res. 2023 Jul;16(7):1450-1461. doi: 10.1002/aur.2969. Epub 2023 Jun 26. PMID 37357811
- See also: Initial Fit Families Program Study — https://clinicaltrials.gov/ct2/show/NCT04612647